CLINICAL TRIAL: NCT00105677
Title: Reasons for Disparities in Joint Replacement Utilization
Brief Title: Understanding the Differences in the Management of Patients With Arthritis of the Knee or Hip
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: ECV 03-201
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2006-10

CONDITIONS: Osteoarthritis; Arthritis, Degenerative; Osteoarthritis, Hip; Osteoarthritis, Knee
Keywords: Racial/ethnic health disparities; Attitudes; Osteoarthritis Management; Patient Perceptions
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip; Osteoarthritis, Knee; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
The purpose of this study is to examine cultural and clinical context factors in African-American and white veterans with knee or hip osteoarthritis with a focus on how these factors may be potentially modifiable determinants of willingness to consider joint replacement.

DETAILED DESCRIPTION:
The study focuses on identifying potentially modifiable determinants of patients� willingness to consider joint replacement as a treatment option for osteoarthritis of the knee or hip. This line of research is informed by not only our prior work but also recent studies on health disparities and patient decision-making. Our long-term goal is the development and evaluation of interventions to target these determinants of willingness in order to eliminate ethnic disparities in joint replacement. The study findings will assist in laying the groundwork for the design of such interventions for patients with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic, frequent knee or hip pain based on the National Health And Nutrition Examination Survey
2. Age >50 and <80 (at least 50 but not to exceed 79 years of age)
3. Severe or extreme knee or hip OA on the Western Ontario and McMaster Universities Osteoarthritis Index (i.e., score greater than or equal to 39)

Exclusion Criteria:

1. Prior history of knee or hip joint replacement
2. Terminal illness (i.e., end-stage cancer, CHF, COPD, etc.)
3. Physician-diagnosed inflammatory arthritis
4. Dementia
5. Prosthetic leg

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 980 (Estimated)
Dates: Start 2004-08; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Kent Kwoh, MD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Arizona, United States

REFERENCES:
- [Result] Jones AC, Kwoh CK, Groeneveld PW, Mor M, Geng M, Ibrahim SA. Investigating racial differences in coping with chronic osteoarthritis pain. J Cross Cult Gerontol. 2008 Dec;23(4):339-47. doi: 10.1007/s10823-008-9071-9. PMID 18561011
- [Result] Emejuaiwe N, Jones AC, Ibrahim SA, Kwoh CK. Disparities in joint replacement utilization: a quality of care issue. Clin Exp Rheumatol. 2007 Nov-Dec;25(6 Suppl 47):44-9. PMID 18021506
- [Result] Groeneveld PW, Kwoh CK, Mor MK, Appelt CJ, Geng M, Gutierrez JC, Wessel DS, Ibrahim SA. Racial differences in expectations of joint replacement surgery outcomes. Arthritis Rheum. 2008 May 15;59(5):730-7. doi: 10.1002/art.23565. PMID 18438917
- See also: Click here for more information about this study: Reasons for Disparities in Joint Replacement Utilization — http://www.cherp.org